CLINICAL TRIAL: NCT03027622
Title: The Effects of Active Surveillance Protocol on Long Term Quality of Life in Patints With Mild Pericoronitis
Brief Title: The Effects of Active Surveillance Protocol on Long Term Quality of Life in Patients With Mild Pericoronitis
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cahit UCOK, DDS PhD, clinical professor, Ankara University
Other Study IDs: 3/5-2015
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Pericoronitis
Keywords: quality of life; pericoronitis; third molar
MeSH Terms: conditions — Pericoronitis | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- long term quality of life: to evaluate conservatively managed third molars with mild pericoronitis at first, third and sixth months by using OHIP-14 TR
  Interventions: Behavioral: quality of life in the patients with mild pericoronitis

INTERVENTIONS:
Behavioral: quality of life in the patients with mild pericoronitis — active surviallence by OHIP-14 TR after treatment

SUMMARY:
The complications that could occur during or after the extraction of the mandibular third molar teeth with pericoronitis affect patient's life quality considerably. Various scales are used to reveal how much the life quality of patients is affected this treatment. The aim of this study is to identify the long term life quality of patients through the OHIP-14 TR scale without removing the mandibular third molar teeth with mild pericoronitis.

DETAILED DESCRIPTION:
Increasing the lenght stay in the mouth at a maximum rate and following the patient up after the necessary treatment and information procedures are completed. As a result of clinical and radiographical examinations fifty-five voluntary patients whose average age was 24 and who have semi or fully errupted vertical mandibular third molar teeth with the diagnosis of mild pericoronitis were included in the study.After the patients in the study filled out the form including their contact and demographic data and dental symptomsand completed OHIP-14 TR scale which last about 5 minutes, their curretage and operculectomy treatments were done under local anesthesia. The patients were invited for reexamination on seventh day after the treatment. Also, an active patient follow up about life quality was performed by phone at 1,3,6 month after the treatment using the self -assessment question form and the OHIP-14 TR scale.

ELIGIBILITY:
Inclusion Criteria:

* having the first episode of mild pericoronitis, having a good periodontal health, having an age between 18 and 25 years
* having a diagnosis of pericoronitis of a vertically erupted or semi erupted lower third molar, having no systemic discomfort and being in the ASA I and ASAII

Exclusion Criteria:

* having no lower third molar with a vertical position
* having a systemic discomfort
* having moderate to severe pericoronitis
* having a history antibiotics or NSAIID

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 55 patients diagnosed with pericoronitis affecting third molars
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Total score of OHIP-14 TR at the begining of experiment | first month
  numeric values of OHIP-14 TR

SECONDARY OUTCOMES:
Total score of OHIP-14 TR at third months | third months
  numeric values of OHIP-14 TR
Total score of OHIP-14 TR at sixth months | sixth months
  numeric values of OHIP-14 TR

IPD SHARING:
Plan to Share IPD: Undecided